CLINICAL TRIAL: NCT05209919
Title: Echocardiographic Assessment and CLInical imPlication of Functional tricuSpid rEgurgitation in Heart Failure With Reduced or Preserved Ejection Fraction (ECLIPSE-HF)
Brief Title: Echocardiographic Assessment and CLInical imPlication of Functional tricuSpid rEgurgitation in Heart Failure With Reduced or Preserved Ejection Fraction
Acronym: ECLIPSE-HF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Collaborators: Cardarelli Hospital (Other); Fondazione C.N.R./Regione Toscana "G. Monasterio", Pisa, Italy (Other Government); Monaldi Hospital (Other); Federico II University (Other); Cava de Tirreni Costiera Amalfitana Hospital Salerno (Unknown); Umberto I Hospital, Nocera Inferiore (Other); Azienda Ospedaliera OO.RR. S. Giovanni di Dio e Ruggi D'Aragona (Other); Azienda Ospedaliera S. Maria della Misericordia (Other); University of Pisa (Other); Niguarda Hospital (Other); IRCCS Policlinico S. Donato (Other); University of Parma (Other); University of Siena (Other); Foligno Hospital (Other); University of Targu Mures, Romania (Other); Szeged University (Other); National Cardiology Hospital, Bulgaria (Other); Bieganski Hospital Lodz, Poland (Unknown); Departement of clinical sciences, Lund University and Skane University Hospidal, Lund Sweden (Unknown); King Faisal Specialist Hospital & Research Center (Other); Piedmont Heart Institute, Inc., Atlanta, GA (Industry); Jewish General Hospital (Other); Ospedali Riuniti di Foggia (Other)
Responsible Party: Principal Investigator, Stefano Ghio, MD, Fondazione IRCCS Policlinico San Matteo di Pavia
Other Study IDs: 0099915/21
Record Dates: First submitted 2021-12-17; First posted 2022-01-27 (Actual); Last update posted 2022-01-27 (Actual); Status verified 2022-01

CONDITIONS: Functional Tricuspid Regurgitation
Keywords: tricuspid regurgitation; heart failure
MeSH Terms: conditions — Tricuspid Valve Insufficiency; Heart Failure | interventions — Echocardiography; Physical Examination; Electrocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Pulmonary arterial hypertension: All patients with pulmonary arterial hypertension and significant functional tricuspid regurgitation
  Interventions: Diagnostic Test: Transthoracic Echocardiography
- HFrEF: All patients with HFrEF and significant functional tricuspid regurgitation
  Interventions: Diagnostic Test: Transthoracic Echocardiography
- HFpEF: All patients with HFpEF and significant functional tricuspid regurgitation
  Interventions: Diagnostic Test: Transthoracic Echocardiography
- Heart Failure mildly-reduced ejection fraction: All patients with Heart Failure mildly-reduced ejection fraction and significant functional tricuspid regurgitation
  Interventions: Diagnostic Test: Transthoracic Echocardiography

INTERVENTIONS:
Diagnostic Test: Transthoracic Echocardiography — All patients undergo physical examination, ECG, Transthoracic Echocardiography, six minutes walking test and blood sample (natruretic peptides, renal and liver function)
  Other Names: six minutes walking test; Physical Examination; 12-lead electrocardiogram; blood sample test

SUMMARY:
Purpose Functional tricuspid regurgitation (FTR) has been shown to be associated with increased morbidity and mortality in several clinical conditions, including heart failure (HF) with reduced left ventricular ejection fraction as well as pulmonary arterial hypertension (PAH). We have designed a study aiming at: characterizing the echocardiographic morphology of the tricuspid valve apparatus and the pathophysiology of FTR in heart failure with reduced, mid-range or preserved left ventricular ejection fraction (HFrEF, HFmrEF, HFpEF) and in PAH patients; correlating the morphologic characteristics of tricuspid valve apparatus with hemodynamic severity of FTR; correlating the severity of FTR with the clinical condition and outcome. Methods The study will be a non-interventional, prospective, international, multicenter, longitudinal study. The minimum number of patients which are expected to be enrolled is 300 HF patients, including HFrEF, HFmrEF and HFpEF patients, whereas 100 PAH patients will serve as control. The patients will be enrolled in 20 centers in Europe, North America and Saudi Arabia. The echocardiographic parameters will be analyzed by the local investigators; a quality control committee will evaluate all data entered in the database to identify potential outliers and a random sample of 10% of cases will be blindly re-analysed in a central core-lab. Conclusions This study has been designed to improve our understanding of pathophysiological mechanisms and clinical relevance of FTR across all HF phenotypes. The results could potentially allow a more appropriate selection of heart failure patients with FTR for tricuspid valve intervention by percutaneous or surgical repair or replacement.

ELIGIBILITY:
Inclusion Criteria:

* consecutive consenting outpatients with HFrEF, HFmrHF, HFpEF or PAH,
* ambulatory visit routinely planned with an echocardiographic examination,
* at the time of the visit at least moderate FTR diagnosed at echocardiography (by visual assessment),
* aged ≥ 18 years old,
* capable to sign an informed consent.

Exclusion Criteria:

* age < 18 years old,
* congenital heart disease,
* heart failure due to organic mitral or aortic valve disease. No examination will be performed in addition to what is routinely planned for patients' evaluation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients to be enrolled are 300 with heart failure and 100 with PAH, given that each center guarantees the enrollment of a minimum number of 20 patients.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2021-11-11 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Time to all-cause death or to first HF hospitalization | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation IRCCS SanMatteo Hospital, Pavia, PV, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ghio S, Bossone E, Mercurio V, Rudski L, Vannan M; RIGHT-NET Investigators. Echocardiographic assessment and clinical implication of functional tricuspid regurgitation in heart failure with reduced or preserved ejection fraction (ECLIPSE-HF) : Rationale and design of the study. Int J Cardiovasc Imaging. 2022 Dec;38(12):2581-2591. doi: 10.1007/s10554-022-02599-8. Epub 2022 Aug 8. PMID 36445668